CLINICAL TRIAL: NCT06532916
Title: Color Stability and Wear Resistance of Direct Flowable and Preheated Resin Composite Veneers Using the Injectable Resin Technique: A Randomized Controlled Clinical Trial.
Brief Title: Color Stability and Wear Resistance of Direct Flowable and Preheated Composite Using the Injectable Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ghada Maghaireh, Dr., King Abdullah University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 751-2023
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Resin Composite Restorations; Esthetic Restorations
Keywords: Resin composites; Injectable resins; Preheated resins

STUDY DESIGN:
Intervention Model Description: The design of the study will be a double blinded (Evaluator and Patient) split-mouth randomized clinical study with two study groups.
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants will be informed about the nature and objectives of the study; however, they will not be informed about the material they are going to receive. The evaluator will not be aware of the treatment groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental)
  Interventions: Other: Experimental: Group1: Estelite Sigma Quick; Other: Experimental: Group 2: Estelite Flow Quick
- Group 2 (Experimental)
  Interventions: Other: Experimental: Group1: Estelite Sigma Quick; Other: Experimental: Group 2: Estelite Flow Quick

INTERVENTIONS:
Other: Experimental: Group1: Estelite Sigma Quick — Preheated conventional composite (Estelite Sigma Quick, Tokuyama Dental Corp, Tokyo, Japan). Estelite Sigma Quick is a resin composite with the following composition (Silica-zirconiasupra-nano, monodispersingc spherica, Bis-GMA, UDMA, TEGDMA).
Other: Experimental: Group 2: Estelite Flow Quick — Second group: Injectable flowable (Estelite Flow Quick, Tokuyama Dental Corp, Tokyo, Japan). Estelite Flow Quick is a resin composite with the following composition (Silica-zirconia, supra-nano monodispersing spherical, Bis-GMA, UDMA,TEGDMA).

SUMMARY:
The aim of this study is to conduct the first clinical trial to assess the color stability and wear resistance of the highly filled injectable flowable composite materials compared to preheated conventional ones and evaluate the in vivo performance of the injectable composite technique.

DETAILED DESCRIPTION:
The design of study will be a modified split-mouth randomized clinical trial with two study groups. 20 patients will be recruited with the need of at least 6 anterior aesthetic restorations. A total of 142 restorations will be assigned into two groups. In the first group, 71 anterior teeth will be restored with flowable composite veneer restorations, and the second group 71 anterior teeth will be restored with heated composite veneer restorations. Both treatment groups will be done using the injectable resin technique. The following parameters will be evaluated at baseline, 6 months and 12 months of clinical service. Color stability will be evaluated using the Vita classical shade guide and a spectrophotometer. Wear resistance will be evaluated by measuring the volumetric material loss through superimposition of images taken at each follow up on baseline images taken by scanning of gypsum replicas using a 3D laser scanner. Clinical performance will be evaluated using the USPHS criteria. It is expected that the color stability, wear resistance and clinical performance of the heated composite restorations will be superior to the flowable restorations.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Asymptomatic sound anterior teeth, or localized Class III/IV/V cavity or restoration
* Patients with irregular tooth anatomies, misalignments, spacing, mild staining, cervical wear that are indicated for direct composite veneers
* Restorations in functional occlusions with an opposing natural tooth.
* Two proximal contacts area with neighboring teeth

Exclusion Criteria:

* Patients with contra-indications for regular dental treatment based on their medical history.
* Patients at a high risk of caries.
* Patients with poor oral hygiene.
* Teeth with compromised periodontal status.
* Evidence of active parafunctional habits or excessive tooth wear.
* Severe discoloration
* Heavy smokers
* Patients with special aesthetic requirements that could not be solved by direct composite veneers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2014-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
The wear resistance of the injectable flowable composite veneers compared to their preheated resin composites counterparts. | Assessment at baseline, 6 months and 1 year after the restorations of the teeth.
  Participants will be assessed at baseline, directly after the finishing and polishing procedure, and at review visits according to the following criteria:
  -The gypsum replicas will be scanned three-dimensionally using a 3D laser scanner at baseline, 6 months and 12 months of clinical service, to analyse the volumetric material loss, which can be associated with structural wear, using 3D analysis software (Medit Link, Medit, Seoul, Republic of Korea) [28, 29] [30] [31] [32]. Follow up images will be superimposed on baseline images
The color stability of the injectable flowable composite veneers compared to their preheated resin counterparts. | Assessment at baseline, 6 months and 1 year after the restorations of the teeth.
  -Shade measurements will be taken at baseline, one week, one month, 3 months and 6 months using the following methods:
  1. Using a spectrophotometer (VITA Easyshade V; VITA Zahnfabrik, Bad Säckingen, Germany), color values (L*, a*, b*) according to the Commission Internationale d'Eclairage (CIELab) will be taken at the middle of each restored tooth using a customized jig to fix the position and in the afternoon with sunlight and standardized room illumination and at each evaluation period. The color changes will be determined using the CIEDE2000 formula.
  2. Using Vita classical shade guide (Vita Zahnfabrik, Bad Säckingen, Germany) and a professional photograph before treatment, at baseline and at each review visit.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A Maghaireh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan